CLINICAL TRIAL: NCT02319863
Title: A Simple Technique of Rapid Ligating the Corresponding Inflow and Outflow Vessels Without Hilus Dissection During Hepatectomy
Brief Title: Rapid Ligating the Corresponding Inflow and Outflow Vessels Without Hilus Dissection During Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chenxp5; 2012ZX10002016-004 (Other Grant/Funding Number: State key project on inflectional disease of China)
Record Dates: First submitted 2014-12-11; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Cancer Progression
Keywords: hepatocellular carcinoma; prognosis
MeSH Terms: conditions — Disease Progression; Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional resection (Active Comparator): Perform hepatectomy with conventional method for HCC patients.
  Interventions: Procedure: hepatectomy (conventional method)
- new method (Experimental): The new technique of rapid ligating the corresponding inflow and outflow vessels without hills dissection before parenchyma transection during hepatectomy.
  Interventions: Procedure: hepatectomy (rapid ligating)

INTERVENTIONS:
Procedure: hepatectomy (conventional method) — A Simple Technique of Rapid Ligating the Corresponding Inflow and Outflow Vessels Without Hilus Dissection During Hepatectomy
  Other Names: liver resection
  Arms: conventional resection
Procedure: hepatectomy (rapid ligating)
  Arms: new method

SUMMARY:
This study examines the role of this simple technique on postoperative metastasis and long term survival.

DETAILED DESCRIPTION:
The only hope of long-term survival for patients with primary hepatocellular carcinoma (HCC) is surgical resection or liver transplantation, the former of which is more feasible at present. However, postoperative recurrence or metastasis is an ominous feature for this disease. Innovation of the surgical procedure for improving prognosis is under emergency request. This study examines the role of this simple technique on postoperative metastasis and long term survival.

During the past 20 years, more 600 patients with primary HCC were performed hepatectomy with the new hemorrhage control technique, and prospective randomized controlled trial (RCT) was applied. We further applied a mice model ligating the pedicle of the lesion-located hepatic lobe before hepatectomy to imitate the clinic practice, and evaluated the role of the new technique on postoperative metastasis and survival.

ELIGIBILITY:
Inclusion Criteria:

* HCC patients who will perform left- or right- hemihepatectomy.

Exclusion Criteria:

1. contraindication for hepatectomy, including gastrointestinal hemorrhage, severe hemorrhagic disorders, explicit acute nonspecific infectious lesion, overt ascites, Child-Pugh Score C,indocyanine green retention rate at 15min (ICGR15)>30%,serum hepatitis B virus (HBV)-DNA>106 copies/ml and serum alanine aminotransferase (ALT)>2×ULN, serum triglycerides>2.0 mmol/L, circulatory shock, stroke, acute myocardial infarction, renal failure, coma of unknown cause;
2. pregnancy;
3. age of<18y or>65y

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 1994-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
recurrence | 12 months
  to examine if there is intrahepatic recurrence
metastasis | 12 months
  to examine if there is intrahepatic metastasis and metastasis in distant organs
mortality | 1 month
  intraoperative death， and death in one month after surgery

SECONDARY OUTCOMES:
Prognosis | 5 years
  to check the 5 years overall survival (OS) and disease free survival (DFS)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, M.D., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Chen XP, Qiu FZ. A simple technique ligating the corresponding inflow and outflow vessels during anatomical left hepatectomy. Langenbecks Arch Surg. 2008 Mar;393(2):227-30; discussion 231-4. doi: 10.1007/s00423-007-0224-z. Epub 2007 Nov 3. PMID 17978838